CLINICAL TRIAL: NCT04041583
Title: Clinical and Radiological Outcomes of Posterior Cervical Fusion Supplemented With Interfacet Spacers
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Andrew Grossbach, Principal Investigator, Assistant Clinical Professor, Ohio State University
Other Study IDs: 2019H0015
Record Dates: First submitted 2019-07-23; First posted 2019-08-01 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cervical Fusion
MeSH Terms: conditions — Klippel-Feil Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Arm 1: Patients undergoing posterior cervical arthrodesis procedures for spondylosis supplemented with CIS involving three or more segmental levels in the subaxial cervicothoracic spine (between C2-upper thoracic)
  Interventions: Device: Cervical Interfacet Spacers

INTERVENTIONS:
Device: Cervical Interfacet Spacers — The use of Cervical Interfacet Spacers is a relatively novel technique shown to be useful for posterior fusion to address symptomatic pseudoarthrosis (fusion failure) after anterior cervical arthrodesis [2]. CIS have a relatively large osteoconductive surface area and are placed under tension in the interfacet space, which together favorably influence bony fusion [2].
  Other Names: (CIS; CORNERSTONE Facet MicroGrafts, Medtronic, Minneapolis, MN)

SUMMARY:
This is a prospective study to assess fusion rates and cervical sagittal parameters following posterior cervical arthrodesis procedures supplemented with CIS. Data will be collected from medical records for up to 730 days after surgery. Data to be collected will be demographic, preoperative clinical information, surgical details, and radiographic information. Patients will also undergo a non-standard of care CT scan 2 years after surgery.

DETAILED DESCRIPTION:
Background and Rationale

Posterior cervical fusion surgeries are performed for degenerative cervical conditions, cervical deformity, cervical tumors, and cervical trauma. They are preferred over an anterior approach when the pathology is located posterior to the spinal cord or when multiple levels must be addressed. Degenerative cervical spondylosis contributes to loss of disc height, facet arthropathy and hypertrophy, and retrolisthesis of the vertebral bodies, all of which can lead to foraminal stenosis, or narrowing around the exiting nerve roots. This is often accompanied by loss of cervical lordosis. During a posterior fusion operation, the restoration of cervical lordosis can worsen this foraminal stenosis and lead to iatrogenic radiculopathy with and estimated incidence between 2.4-50%. Cadaveric studies have shown the insertion of interfacet spacers in the cervical spine increase foraminal height, and serve to indirectly decompress the exiting nerve roots. Another common complication of cervical spine surgery is C5 palsy, which has been reported in 4.6% of patient undergoing posterior cervical spine decompressive procedures, including decompression and fusion. Patients suffering from iatrogenic C5 palsy have significantly increased recovery times, and often require additional services such as imaging studies (CT, MRI) and increased need for physical and occupational therapy, thus increasing costs. Given the ability to decompress the neuroforamen with interfacet spacers, they could potentially be an effective technique for reducing the incidence of C5 palsy.

The use of cervical interfacet spacers (CIS; CORNERSTONE Facet MicroGrafts, Medtronic, Minneapolis, MN) is a relatively novel technique shown to be useful for posterior fusion to address symptomatic pseudoarthrosis (fusion failure) after anterior cervical arthrodesis. CIS have a relatively large osteoconductive surface area and are placed under tension in the interfacet space, which together favorably influence bony fusion. Current techniques for posterior cervical fusion rely on graft placement using bone extenders placed in the posterolateral space, which is not under a compressive load. Wolfe's law dictates that certain amounts of loading of bone grafts is required to achieve bony fusion. Therefore, the use of CIS could potentially increase fusion rates after posterior cervical arthrodesis procedures and reduce or eliminate the need for use of bone graft extenders. Reassuringly, radiologic studies have shown that despite the increase in foraminal height, the use of CIS does not lead to loss of cervical lordosis.

Study Objective

To date, there have been no prospective studies examining the use of cervical interfacet spacers. The investigators propose to undertake a prospective study to assess fusion rates and cervical sagittal parameters following posterior cervical arthrodesis procedures supplemented with CIS.

Primary Outcome Measures The primary outcome measures will include (i) the rate of cervical fusion measured on post-operative radiographs and CT scans performed at 2-years and (ii) cervical sagittal alignment parameters as measured on post-operative radiographs.

Secondary Outcome Measures The secondary outcome measures will include post-operative patient reported outcomes including NRS, NDI, and SF-36 RAND. As well, all neurological adverse events will be prospectively collected.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Symptomatic multi-level degenerative spondylosis necessitating posterior cervical arthrodesis in the subaxial cervicothoracic spine (between C2-upper thoracic).
* Surgery performed within the Department of Neurological Surgery at The Ohio State University Wexner Medical Center (OSUWMC)

Exclusion Criteria:

* Traumatic injury
* Co-morbidity requiring medication use that may interfere with bone or soft tissue healing (i.e., high dose oral or parenteral glucocorticoids, immunosuppressive agents, methotrexate) - at discretion of investigator
* Severe co-morbidities (e.g., heart, respiratory, or renal disease)
* Recent (<3 yrs) or co-incident spinal tumor or infection
* Concurrent involvement in another investigational drug or device study that could confound study data
* History of substance abuse (recreational drugs, prescription drugs or alcohol) that could interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up
* Subjects who are pregnant or plan to become pregnant in the next 24 months
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing posterior cervical arthrodesis procedures for spondylosis supplemented with CIS involving three or more segmental levels in the subaxial cervicothoracic spine (between C2-upper thoracic)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Cervical Fusion | 2-Years
  Cervical Fusion Measured on Post-Operative Radiographs and CT scans
Cervical Sagittal Alignment Parameters | 2-Years
  Cervical Sagittal Alignment Parameters measured on post-operative radiographs

SECONDARY OUTCOMES:
NRS | 2-Years
  Numerical Rating Score for Pain from 0-10 where lower values represent a better outcome
NDI | 2-Years
  Neck Disability Index from 0-100% where lower values represent a better outcome
SF-36 RAND | 2-Years
  Quality of Life Measures from 0-100 where higher values represent a better outcome
Neurological Adverse Events | 2-Years
  Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Grossbach, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan LA, Gerard CS, Anderson PA, Traynelis VC. Effect of machined interfacet allograft spacers on cervical foraminal height and area. J Neurosurg Spine. 2014 Feb;20(2):178-82. doi: 10.3171/2013.11.SPINE131. Epub 2013 Dec 13. PMID 24328759
- [Result] Kasliwal MK, Corley JA, Traynelis VC. Posterior Cervical Fusion Using Cervical Interfacet Spacers in Patients With Symptomatic Cervical Pseudarthrosis. Neurosurgery. 2016 May;78(5):661-8. doi: 10.1227/NEU.0000000000001087. PMID 26516824
- [Result] Mummaneni PV, Meyer SA, Wu JC. Biological approaches to spinal instrumentation and fusion in spinal deformity surgery. Clin Neurosurg. 2011;58:110-6. doi: 10.1227/neu.0b013e3182270009. No abstract available. PMID 21916134
- [Result] Tan LA, Straus DC, Traynelis VC. Cervical interfacet spacers and maintenance of cervical lordosis. J Neurosurg Spine. 2015 May;22(5):466-9. doi: 10.3171/2014.10.SPINE14192. Epub 2015 Feb 13. PMID 25679233
- [Result] Fogel GR, Toohey JS, Neidre A, Brantigan JW. Fusion assessment of posterior lumbar interbody fusion using radiolucent cages: X-ray films and helical computed tomography scans compared with surgical exploration of fusion. Spine J. 2008 Jul-Aug;8(4):570-7. doi: 10.1016/j.spinee.2007.03.013. Epub 2007 May 29. PMID 17544854
- [Result] Turel MK, Kerolus MG, Traynelis VC. Machined cervical interfacet allograft spacers for the management of atlantoaxial instability. J Craniovertebr Junction Spine. 2017 Oct-Dec;8(4):332-337. doi: 10.4103/jcvjs.JCVJS_87_17. PMID 29403245

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT04041583/Prot_SAP_000.pdf